CLINICAL TRIAL: NCT07372820
Title: METAB-HTX: Prospective, Longitudinal Cohort Study Evaluationg Cardiac and Systemic Metabolism After Heart Transplantation
Brief Title: METABolic Deterioration in HTX Determines Outcomes
Acronym: METAB-HTX
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: METAB-HTX
Record Dates: First submitted 2025-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation
Keywords: cardiac metabolism; Systemic Metabolism; cardiac function; heart transplant; heart failure; Type 2 diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples:including circulating citrullinated histone H3 (H3cit)-DNA complexes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Adult advanced heart failure patients listed for HTx: Patients with advanced heat failure (AHF) and listed for heart transplantation (HTx)

SUMMARY:
METAB-HTX is a prospective, longitudinal cohort study evaluating cardiac and systemic metabolism in heart transplant recipients.

DETAILED DESCRIPTION:
Bankground:

Heart Transplantation (HTS) is the treatment of choice for advanced heart failure, yet long-time survival rates require further improvement. Recent studies highlight obesity, type 2 diabetes, renal dysfunction, and hepatic impairment as key contributors to post-transplant mortality. Furthermore, critical questions persist in understanding the optimal metabolic surveillance post-HTX, the direct association between metabolic dysregulation and cardiac dysfunction, inter-organ interactions linking metabolic decline to hepatic/renal impairment and the timing of therapeutic strategies.

Therefore: METAB-HTX study aims to address these open questions, hypothesizing that metabolic deterioration post-HTX is associated with impaired cardiac function and survival.

Study Design:

The study employs advanced multi-modal phenotyping to investigate interactions between cardiac function, metabolic dysregulation, and systemic organ dysfunction.

Cardiac Phenotyping:

* Imaging: Serial echocardiography, cardiac MRI (cMRI), and magnetic resonance spectroscopy (MRS) for myocardial structure, perfusion, and metabolic profiling.
* Vascular Evaluation: Coronary angiography to detect macro- and microvascular coronary allograft vasculopathy (CAV).
* Rejection Monitoring: Protocol-driven endomyocardial biopsies for histopathological grading.

Metabolic phenotyping:

* Serial oral glucose tolerance tests, homeostasis model assessment, type 2 diabetes endotyping and muscle biopsies.
* Advanced lipid panels, HDL functional assays and plasma membrane lipid fluidity analyses.
* MRI/MRS-based quantification of adipose tissue distribution and ectopic fat deposition.

Systemic Organ Evaluation:

* renal and liver function.

Molecular and Multi-Omics Integration:

* Myocardial Energy Metabolism, Genomic/Transcriptomic Profiling, Thromoboinflammation and Neoplasia Risk.

This innovative study aims to bridge critical gaps in understanding post-transplant metabolic pathophysiology, potentially refining surveillance protocols and guiding targeted therapies to improve long-term survival through precision medicine strategies

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Planned or already conducted heart transplantation
* Informed consent

Exclusion Criteria:

* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the heart transplant waiting list, as well as post-heart transplantation
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
diastolic and systolic left ventricular function | Baseline, 1 year, and 2 years after heart transplantation
  in cardiac MRI or echocardiography
CAV diagnosis | Baseline, 1 year, and up to 24 months
  coronary angiography, intravascular imaging and intravascular physiology measuraments
Allograft rejection will be evaluated by endomyocardial biopsy | 1 year and 5 years after heart transplantation
  Tissue specimens will be collected from the interventricular septum and analyzed by cardiac transplant pathologists. Myocardial inflammation will be assessed in endomyocardial biopsies using immunohistochemistry followed by quantitative digital image analysis. Inflammatory cell infiltration will be quantified as the number of positive cells per square millimeter (mm²), providing a quantitative measure of myocardial inflammatory burden. In addition, biopsy tissue will be used for exploratory molecular analyses.
Worsening of kidney function | Baseline, 1 year, and 2 years after heart transplantation
  Renal function will be assessed using estimated glomerular filtration rate (eGFR) as the primary quantitative measure. eGFR will be calculated from serum creatinine and cystatin C obtained from periodic blood sampling. Additional renal assessments, including duplex sonography, urinary markers, and immunological parameters, will be used for supportive and exploratory analyses.
Infection requiring heath care professional interventions | Baseline, 1 year, and 2 years after heart transplantation
  clinical events, labs (CRP) , outpatient contact, hospitalisation.
Diagnosis of malignencies | Baseline, 1 year, and 2 years after heart transplantation
  By whole-body CT scans, screening for occult blood within the stool and if indicated gastroscopy and coloscopy. Analysis of epigenetic alterations in leukocytes which are associated with post HTX events like neoplasia.
Worsening of metabolic derangements | Baseline, 1 year, and 2 years after heart transplantation
  Changes in glucose and lipid metabolism, insulin resistance, HDL function, and body fat distribution will be assessed using blood tests, oral glucose tolerance, and imaging in selected participants.
Liver deterioration | Baseline, 1 year, and 2 years after heart transplantation
  Liver structure and function will be assessed using blood tests (liver enzymes, bilirubin, albumin, INR), imaging (ultrasound, CT, transient elastography), and fibrosis scores (FIB-4) in selected participants.

SECONDARY OUTCOMES:
Hospitalisation due to heart transplant events | up to 5 years (follow-up in clinical routine)
  Number of hospitalisations due to heart transplant-related events after study inclusion
Cardiovascular mortality and all-cause mortality | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
Re-transplantation or ventricular assist device implantation | Through study completion, up to 5 years after heart transplantation
  Incidence of re-transplantation or ventricular assist device implantation during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic of Cardiology, Pneumology and Vascular Medicine at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pneumology and Angiology, Düsseldorf, North Rhine-Westphalia, Germany